CLINICAL TRIAL: NCT02832531
Title: INVestIgation of rheumatiC AF Treatment Using Vitamin K Antagonists, Rivaroxaban or Aspirin Studies
Brief Title: INVestIgation of rheumatiC AF Treatment Using Vitamin K Antagonists, Rivaroxaban or Aspirin Studies, Superiority
Acronym: INVICTUS-ASA
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Focus on recruitment for non-inferiority trial
Sponsor: Population Health Research Institute (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INVICTUS - ASA
Record Dates: First submitted 2016-01-07; First posted 2016-07-14 (Estimated); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Rheumatic Heart Disease
Keywords: atrial fibrillation; stroke
MeSH Terms: conditions — Rheumatic Heart Disease; Atrial Fibrillation; Stroke | interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (15 mg) (Experimental): Rivaroxaban 15 mg od (n ~ 1000)
  Interventions: Drug: Rivaroxaban (15 mg)
- Aspirin (ASA) (Active Comparator): Aspirin 100 mg od (n~1000)
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Rivaroxaban (15 mg) — Rivaroxaban is superior to aspirin for the prevention of the composite of stroke or systemic embolism in patients with RVHD with AF or flutter who are unsuitable for VKA therapy, or in patients with RVHD without AF or Flutter with at least one of the following:
  1. Left atrial enlargement ≥ 5.5 cm, OR
  2. Left atrial spontaneous echo contrast OR
  3. Left atrial thrombus OR
  4. Frequent ectopic atrial activity (>1000/24 hours) on Holter ECG.
  Other Names: Xarelto
  Arms: Rivaroxaban (15 mg)
Drug: Aspirin — Rivaroxaban is superior to aspirin for the prevention of the composite of stroke or systemic embolism in patients with RVHD with AF or flutter who are unsuitable for VKA therapy, or in patients with RVHD without AF or Flutter with at least one of the following:
  1. Left atrial enlargement ≥ 5.5 cm, OR
  2. Left atrial spontaneous echo contrast OR
  3. Left atrial thrombus OR
  4. Frequent ectopic atrial activity (>1000/24 hours) on Holter ECG.
  Other Names: acetylsalicylic acid
  Arms: Aspirin (ASA)

SUMMARY:
This program is a comprehensive evaluation of rheumatic valvular heart disease (RVHD), Atrial fibrillation (AF)/flutter and stroke.

A prospective, randomized, open-label superiority trial comparing rivaroxaban to aspirin in high risk patients either with AF and unsuitable for VKA or without AF and with high risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. RVHD diagnosed by echocardiography at any time prior to enrollment
2. Age ≥18
3. Increased risk of stroke by any of the following

   1. CHA2DS2-VASc score ≥ 2 OR
   2. Moderate/Severe mitral stenosis with valve area ≤2.0 cm2 OR
   3. Left atrial spontaneous echo contrast OR
   4. Left atrial thrombus
4. Heart Rhythm

   1. AF or Flutter and unsuitable for VKA therapy. (AF or Flutter should be documented on baseline 12-lead ECG, or on a previous 12-lead ECG, Holter monitor, in-hospital ECG rhythm strip or Pacemaker or ICD electrogram). OR
   2. In the absence of AF or Flutter, patients would be eligible in the presence of any one of the following:

   <!-- -->

   1. Left atrial enlargement ≥5.5 cm OR
   2. Left atrial spontaneous echo contrast OR
   3. Left atrial thrombus OR
   4. Frequent ectopic atrial activity (>1000/24 hours) on Holter monitoring

Exclusion Criteria:

1. Refusal to give informed consent
2. Actively involved in any study that would compromise the protocol of INVICTUS Trial
3. Severe co-morbid condition with life expectancy < 1 year
4. Other serious condition(s) or logistic factors likely to interfere with study participation or with the ability to complete the trial, as appropriate to country or region.
5. Likely to have valve replacement surgery within 6 months
6. Mechanical valve prosthesis or other condition requiring treatment with VKAs. Patients with deep vein thrombosis or recent pulmonary embolism can be enrolled where both VKAs and rivaroxaban are approved.
7. Contraindication to the study medication of the trial

   * Allergy to rivaroxaban
   * Allergy to VKAs ( non-inferiority trial)
   * Allergy to aspirin ( superiority trial)
8. Severe renal insufficiency with an calculated creatinine clearance (Cockcroft-Gault) <15 ml/min
9. Serious bleeding in the past six months or at high risk for bleeding
10. Moderate to severe hepatic impairment
11. Ongoing need for dual antiplatelet therapy (patients with on-going aspirin therapy ≤100 mg per day are not excluded)
12. Ongoing need for dual strong inhibitors of CYP-3a4 or p-glycoprotein inhibitor.
13. Received an investigational drug in the past 30 days
14. Patients considered unsuitable for trial inclusion because of unwillingness to attend follow up visits
15. Women who are pregnant and/or breastfeeding
16. Women of child bearing age who do not use an effective form of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Time from randomization to the first occurrence of Stroke or systemic embolism | Approximately 4 years
  Stroke (Ischemic, hemorrhagic or undetermined type)

SECONDARY OUTCOMES:
Time from randomization to the first occurrence of Myocardial Infarction (MI) | Approximately 4 years
Time from randomization to time of vascular death | Approximately 4 years
  Vascular death includes death due to stroke, myocardial infarction, heart failure or cardiogenic shock, sudden death or any other death due to cardiovascular causes. In addition, death due to hemorrhage will be included

OTHER OUTCOMES:
Time from randomization to the first occurrence of a Major bleed | Approximately 4 years
  Using the International Society on Thrombosis and Haemostasis (ISTH) major bleeding definition

IPD SHARING:
Plan to Share IPD: No
cumulative participant data only